CLINICAL TRIAL: NCT00196430
Title: Prospective, Controlled Three-Armed Study About Effectiveness and Compatibility of Silver-Containing Textiles for Treatment of Acute Neurodermatitis
Brief Title: Study About Effectiveness of Silver-Containing Textiles for Treatment of Acute Neurodermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Julius Zorn GmbH, Aichach, Germany (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: III PV 08/03
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Neurodermatitis
MeSH Terms: conditions — Neurodermatitis | interventions — Adrenal Cortex Hormones

INTERVENTIONS:
Device: silver-contained textiles
Drug: corticosteroid

SUMMARY:
The purpose of this study is to investigate whether the treatment of acute neurodermitis with silver-contained textiles is equivalent or more effective to the conservative exogenous treatment with a corticosteroid. Secondary aim is to define skin comfortability of the textiles.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute Neurodermitis
* Age: 2-70 years
* Patients are mobile
* Patient's information and willingness to participate

Exclusion Criteria:

* Acute viral infection (herpes zoster, eczema herpeticum)
* Acute staphylodermas
* Other skin-diseases affecting outcomes of intervention (e.g. psoriasis)
* Current UV-Treatment
* Current other immunosuppressive or immunomodulated Therapy
* Current antimicrobial Therapy (e.g. antibiotics)
* Severe general diseases (e.g. melanoma, renal insufficiency, autoimmune diseases)
* Pregnancy
* Fertile females without effective contraception

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32
Dates: Start 2004-01; Study Completion 2004-08

PRIMARY OUTCOMES:
SCORAD at days -3,0,7,14,28,56 for every group

SECONDARY OUTCOMES:
Influence of silver containing textiles in reducing bacterial skin colonization (especially Staph. aureus)
Consumption of corticosteroids at days 0-28
Consumption of corticosteroids at days 28-56
Pruritus under textiles
Evaluation of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jünger, Prof. Dr., Principal Investigator — Clinic and Polyclinic of Dermatology, University of Greifswald; Andrea Ladwig, Study Chair — Clinic and Polyclinic of Dermatology, University of Greifswald
Locations (1):
- Clinic and Polyclinic of Dermatology, Ernst-Moritz-Arndt-University of Greifswald, Greifswald, Fleischmannstr. 42-44, Germany